CLINICAL TRIAL: NCT04691817
Title: A Phase Ib-II Trial of Tocilizumab and Atezolizumab in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Refractory to 1st Line Immune Checkpoint Inhibitor-Based Therapy
Brief Title: Tocilizumab and Atezolizumab in Adults With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Refractory to 1st Line Immune Checkpoint Inhibitor-Based Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 16520
Record Dates: First submitted 2020-12-08; First posted 2020-12-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab and Tocilizumab (Experimental): Participants receive Atezolizumab 1200mg IV and Tocilizumab 6mg/kg IV (or Tocilizumab 4mg/kg IV) every 21 days
  Interventions: Drug: Atezolizumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Atezolizumab — 1200mg infusion
  Other Names: Tecentriq
Drug: Tocilizumab — Tocilizumab 6mg/kg or 4mg/kg infusion
  Other Names: Actemra, RoActemra, RO4877533

SUMMARY:
This is a research study to evaluate the safety and effectiveness of tocilizumab in combination with atezolizumab to treat non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced non-squamous NSCLC (Stage IV or recurrent after initial curative intent therapy) in adults age 18 or older
* Prior exposure to at least 1 line of therapy
* Exposure to a including checkpoint inhibitor in line of therapy immediately prior to enrollment on trial
* ECOG PS 0-2

Exclusion Criteria:

* Presence of a driver mutation that is susceptible to targeted therapy
* No greater than CTCAE v5 grade 3 toxicity attributed to prior immunotherapy
* Other active invasive malignancy requiring ongoing therapy
* Evidence of progressing or untreated brain metastases
* Evidence or history of leptomeningeal disease
* Uncontrolled tumor related pain
* History of an autoimmune disease or IPF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From first dose of protocol treatment until radiologic disease assessment at 12 weeks.
  Assess the proportion of patients with a radiologic response by RECIST 1.1 at 12 weeks.

SECONDARY OUTCOMES:
Overall survival (OS) | From first dose of protocol treatment until death due to any cause or last patient contact alive until 3 months after study closure.
  Estimate the time from first dose of protocol treatment until death due to any cause or last patient contact alive until 3 months after study closure
Dose Limiting Toxicities of the combination | From first dose of protocol treatment until 49 days post treatment
  Determine dose limiting toxicities of the combination
Progression free survival (PFS). | From 1st dose of treatment until 1st radiologic disease progression, unequivocal clinical progression, or death due to any cause censored at the last scheduled disease assessment on study if no progression date registered, assessed up to 24 months.
  Estimate the time from first dose of protocol treatment until first radiologic disease progression, unequivocal clinical progression, or death due to any cause censored at the last scheduled disease assessment on study if there is no progression date registered.

OTHER OUTCOMES:
Clinical outcomes | From enrollment until dealth due to any cause or last patient contact alive until 3 months after study closure
  Correlate clinical outcomes with potential markers of immune escape and changes in the tumor microenvironment and blood using a novel field theory based methods under development by Cold Spring Harbor Laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Melina Marmarelis, MD, MSCE, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No